CLINICAL TRIAL: NCT06656585
Title: Evaluation of the Effect of a Food Selectivity Intervention Through Virtual Reality in Children with Autism Spectrum Disorders
Brief Title: Exploring Virtual Reality As an Intervention for Food Selectivity: a Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Fondazione di Comunità Messina onlus (Unknown)
Responsible Party: Principal Investigator, Flavia Marino, Principal Investigator, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2024-011
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; children; food selectivity; virtual reality
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Food selectivity Group (2) (Experimental): 15 children in the comparator group who will undergo the treatment perform the procedure individually using the traditional method.
  Interventions: Other: Traditional food selectivity protocol
- Food selectivity group (1) (Experimental): 15 children in the experimental group who will undergo the treatment perform the procedure individually with exposure to foods through Oculus
  Interventions: Other: Individual food selectivity protocol

INTERVENTIONS:
Other: Individual food selectivity protocol — Children in the experimental group wear Oculus headsets and interact with virtual foods for 20 minutes. In the "Pairing in the Kitchen" phase, Oculus is removed. Two identical plates with 6 foods are placed in front of the child. The operator, seated next to the child, interacts with the food without eating it, maintaining a positive expression, and discussing non-food topics. No prompts to eat are given, and the child can leave at any time. Progress to the next phase if the child sits calmly for 30 seconds across 3 sessions.
  Shaping Phase: Two identical plates are prepared. The operator comments on the food and keeps a small container of the child's favorite food visible but out of reach. Any food-related behavior is reinforced with praise and the favorite food. Target behaviors are adjusted if no response occurs for 15 seconds or if negative emotions are observed. Differential reinforcement is used.
  Arms: Food selectivity group (1)
Other: Traditional food selectivity protocol — Step 1:Pairing in the Kitchen Propose enjoyable activities in the kitchen. Move to Step 2 when the child plays in the kitchen for 5 minutes over 3 consecutive sessions.
  Step 2:Transition to Kitchen Two plates with 6 identical foods are placed in the kitchen. The operator engages the child in a welcome game, waiting 30 seconds for spontaneous interaction. If no response, the operator prompts the child to go to the kitchen. If the child doesn't follow within 30 seconds, the session is postponed. The operator sits next to the child and interacts with the food, without encouraging the child to eat. Progress when the child stays seated for 30 seconds without problem behavior for 3 sessions.
  Step 3:Shaping Two plates are prepared, and the operator comments on the food. A visible container with the child's favorite food is used for reinforcement. Target behaviors are reinforced with praise and the favorite food. Adjust behaviors if there's no response for 15 seconds or negative emotions occur
  Arms: Food selectivity Group (2)

SUMMARY:
Food selectivity is a common challenge among children with Autism Spectrum Disorder (ASD), with significant impacts on their nutrition and well-being. The main purpose of this study is to promote children's active participation in mealtime routines and encourage experimentation with new foods through an approach that emphasizes joy and serenity during mealtimes. The study will involve children with ASD between the ages of 4 and 10 years, of both sexes. Food selectivity will be assessed through interviews with parents and the use of specially created cards.

The protocol will include 45-minute sessions, twice a week, for a total of 48 sessions. The children will wear an Oculus headset and be exposed to the foods through this virtual reality tool, enhancing their engagement and willingness to try new foods in a fun and immersive way.

ELIGIBILITY:
Inclusion Criteria:

* Food selectivity upon parental referral
* Child with diagnosis of autism

Exclusion Criteria:

* presence of other medical disorders

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-17 (Estimated)

PRIMARY OUTCOMES:
Brief Autism Mealtime Behavior Inventory (BAMBI) | The evaluation sessions will be scheduled pre and post intervention.The test needs approximately 20 minutes to complete for parents. The tests will be scheduled pre intervention and at the study conclusion,about after 6 months.
  the Bambi measures food selectivity, disruptive behavior, food refusal and rigidity at mealtime
  The 18-item Brief Autism Mealtime Behavior Inventory (BAMBI) is a parent-report questionnaire that was created to identify mealtime habits unique to kids with ASD.
  The BAMBI is rated on a Likert scale of 1 to 5, where 1 represents "never" occurring behavior during mealtime and 5 represents "always" occurring behavior. For four of the items that rate constructive mealtime behaviors, reversed scoring is applied. The sum of the 18 elements is used to create the total frequency score, with higher scores indicating more issues with behavior during meals.
Inventory of food preferences | The evaluation sessions will be scheduled pre and post intervention.The test needs approximately 20 minutes to complete for parents. The tests will be scheduled pre intervention and at the study conclusion, about after 6 months.
  The food preference inventory includes a list of foods that is submitted to the parent. Asked how often the food is consumed by the child and family.
General assessment | The evaluation sessions will be scheduled pre and post intervention.The test needs approximately 15 minutes to complete for parents. The tests will be scheduled pre intervention and at the study conclusion,about after 6 months.
  The general assessment includes a personal data sheet, the section relating to nutrition and therefore to the dietary regime, the type of selectivity and dysfunctional behaviours. Finally there is the adaptive functioning card relating to autonomy during meals.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Istituto per la Ricerca e l'Innovazione Biomedica
Locations (1):
- Istituto per la Ricerca e l'Innovazione Biomedica, Messina, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] M. M. Essa, M. W. Qoron!eh (eds.), Personalized Food Intervention and Therapy for Autism Spectrum Disorder Management, Advances in Neurobiology 24, https://doi.org/10.1007/978-3-030-30402-7_26
- [Background] Banire B, Khowaja K, Mansoor B, Qaraqe M, Al Thani D. Reality-Based Technologies for Children with Autism Spectrum Disorder: A Recommendation for Food Intake Intervention. Adv Neurobiol. 2020;24:679-693. doi: 10.1007/978-3-030-30402-7_26. PMID 32006380
- [Background] Esposito M, Mirizzi P, Fadda R, Pirollo C, Ricciardi O, Mazza M, Valenti M. Food Selectivity in Children with Autism: Guidelines for Assessment and Clinical Interventions. Int J Environ Res Public Health. 2023 Mar 14;20(6):5092. doi: 10.3390/ijerph20065092. PMID 36982001
- [Background] Peterson KM, Piazza CC, Ibanez VF, Fisher WW. Randomized controlled trial of an applied behavior analytic intervention for food selectivity in children with autism spectrum disorder. J Appl Behav Anal. 2019 Oct;52(4):895-917. doi: 10.1002/jaba.650. PMID 31642526
- [Background] Piazza CC, Patel MR, Santana CM, Goh HL, Delia MD, Lancaster BM. An evaluation of simultaneous and sequential presentation of preferred and nonpreferred food to treat food selectivity. J Appl Behav Anal. 2002 Fall;35(3):259-70. doi: 10.1901/jaba.2002.35-259. PMID 12365739